CLINICAL TRIAL: NCT06724900
Title: A Phase 1/2 Study of KB304, a Replication-Defective, Non-Integrating Vector Expressing Human Type III Collagen (COL3) and Tropoelastin for the Treatment of Wrinkles
Brief Title: A Study Assessing KB304 for the Treatment of Wrinkles in Women
Acronym: Pearl-2
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KB304-01
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-12

CONDITIONS: Wrinkles in Decolletage; Pigmentation; Décolleté Wrinkles
Keywords: Krystal Biotech; wrinkles in decolletage; pigmentation in decolletage; décolleté wrinkles
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KB304 (Experimental)
  Interventions: Biological: KB304
- Placebo (Placebo Comparator)
  Interventions: Drug: 0.9% Normal Saline (NS)

INTERVENTIONS:
Biological: KB304 — Genetically modified herpes simplex type 1 virus
  Arms: KB304
Drug: 0.9% Normal Saline (NS) — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the safety and efficacy of KB304, an investigational gene therapy to correct moderate to severe wrinkles in the décolleté region (V-shaped chest area). KB304 is an investigational gene therapy that delivers functional, full-length human collagen (COL3) and elastin (tropoelastin) to the skin through small injections using the Sponsor's genetically engineered Herpes Simplex Virus (HSV-1) vector. The study is a randomized double-blind study and participants will receive either KB304 (active group) or placebo (inactive group).

ELIGIBILITY:
Inclusion Criteria:

* Female in good general health, as determined by the Investigator, aged ≥18 and ≤75 at the time of consent.
* Presence of moderate to severe dynamic wrinkles in the décolleté Target Area, as determined by the Investigator on the JDWS.
* A Fitzpatrick skin phototype score of I-IV.
* A negative urine pregnancy test at Screening and Day 1 (Visit 2) for subjects of child-bearing potential.
* Signed and dated informed consent and willingness to attend all study visits and complete all procedures required by the protocol.

Exclusion Criteria:

* Any transient or chronic skin condition, disorder, or infection within 20 cm of the Target Area at Day 1 (Visit 2) that, in the opinion of the Investigator, may interfere with the interpretation of study results.
* Scars, tattoos or tanned skin (defined as skin that is tanned from sun exposure, tanning beds, or an applied skin color such as a spray tan) within the Target Area at Day 1 (Visit 2).
* History of laser treatment, microneedling, chemical peels within 3 months of Day 1 (Visit 2), or botulinum toxin within 6 months of Day 1 (Visit 2) to the Target Area.
* History of surgical procedures to Target Area, including removal of benign or malignant skin cancers that, in the opinion of the Investigator, may interfere with the interpretation of study results.
* Administration of a cosmetic and/or investigational agent, in the Target Area within 6 months of Day 1 (Visit 2), that, in the opinion of the Investigator, may interfere with the interpretation of study results.
* Any condition (including a history or current evidence of substance abuse or dependence, ongoing systemic infection, infection local to the Target Area, immunosuppression, or recent history of or active malignancy in the Target Area) that, in the Investigator's opinion, would impact the subject's ability to complete all study-related procedures and/or poses an additional risk to the assessment of safety of the Investigational Product.
* Subject who is pregnant or nursing.
* Subject who is unwilling to comply with contraception requirements per-protocol.
* Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol, in the opinion of the Investigator

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of KB304 versus placebo administered by intradermal injection | Up to 4 months
  Treatment related adverse events as assessed by CTCAE

SECONDARY OUTCOMES:
To evaluate the effect of KB304 versus placebo on dynamic wrinkles of the décolleté area. | Up to 4 months
  Change from baseline as compared to placebo in the Investigator's live assessment (using a 6-Point Global Aesthetic Improvement Scale (GAIS)) and the participants' self-assessment where +2 is much improved and -2 is not applicable.
To evaluate the effect of KB304 versus placebo on dynamic wrinkles of the décolleté area. | Up to 4 months
  Change from baseline as compared to placebo in the Investigator's live assessment (using a 5-Point Jeune Décolleté Wrinkle (JDWS) Photographic Scale) where 0 is none and 4 is extremely severe.
To evaluate the effect of KB304 versus placebo on dynamic wrinkles of the décolleté area. | Up to 4 months
  Change from baseline as compared to placebo in subject satisfaction using a 6-Point Scale where +2 is very satisfied and -2 is not applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Steve Yoelin Medical Associates, Newport Beach, California, United States